CLINICAL TRIAL: NCT02243670
Title: Feasibility and Validity of Using a Novel Artificial Intelligence Platform to Monitor and Optimize Medication Adherence in Patients Receiving Opioid Replacement Therapy
Brief Title: Using Artificial Intelligence To Monitor Medication Adherence in Opioid Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AiCure (Industry)
Collaborators: Orexo AB (Industry); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIC-HHSN271201300036C-01; HHSN271201300036C (Other: NIDA Contract)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Opiate Addiction; Medication Non-adherence; Addiction; Opioid Dependence
Keywords: opioid addiction; opioid substitution therapy; addiction; buprenorphine maintenance treatment; opioid dependence; substitution treatment; noncompliance; opiate addiction; Zubzolv® maintenance; adherence monitoring; directly observed therapy; medication adherence; adherence; mobile; electronic monitoring; wireless; mobile device; artificial intelligence; facial recognition; computer vision; visual confirmation; sublingual buprenorphine/naloxone; nonadherence
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence; Behavior, Addictive; Patient Compliance; Directly Observed Therapy | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AiCure monitoring and intervention (Experimental): Participants will use the AiCure app to monitor ingestion of all prescribed doses of Zubsolv®.
  Interventions: Device: AiCure monitoring and intervention

INTERVENTIONS:
Device: AiCure monitoring and intervention — Participants will use the AiCure app to monitor ingestion of all prescribed doses of Zubsolv®. If a participant misses a dose, takes an incorrect dose, or their data are flagged for suspicious activity, they will be contacted by research staff or the AiCure study team through automated SMS text or by phone.
  Other Names: Automated DOT

SUMMARY:
This study uses an artificial intelligence platform to automatically confirm medication ingestion. The Health Insurance Portability and Accountability Act (HIPAA)-compliant platform can be downloaded as an 'app' onto any smartphone to automate directly observed therapy (Automated DOT®). Real-time patient adherence data are encrypted and automatically sent to a centralized web-based dashboard for use by healthcare professionals or research staff. Unlike Facetime® or Skype®, the system relies on computer vision algorithms to confirm the process of medication administration; no human review is necessary.

The purpose of this study is to evaluate the feasibility and acceptability, and measure the accuracy, of the AiCure platform ("platform") in patients being treated for opioid dependence with Zubsolv® over the course of 12 weeks. The following aims will be tested: 1) to assess the feasibility and acceptability to both participants and study staff in using AiCure to monitor medication adherence; 2) to evaluate the acceptability of using AiCure to optimize care pathways; and 3) to measure the reliability and validity of AiCure in detecting interruptions in treatment. To assess feasibility and acceptability of the platform, we will measure rates of physician satisfaction and user acceptance. Optimization of care pathways will be measured by assessing the sustainability of AiCure use over 12 weeks (retention rates) and measuring illicit opioid use (urine drug screens) compared to historical data. Reliability and validity of AiCure will be measured by comparing AiCure adherence against pharmacokinetic data.

All participants will be requested to take each of their prescribed doses using the app. Participants will be able to download the app onto their own smartphone or will be provisioned a device at the start of the study. The data captured during the medication ingestion process will be automatically encrypted and stored on the participant smartphone and uploaded wirelessly to a cloud-based dashboard. If a participant is non-adherent (missed dose, incorrect dosage) or if suspicious behavior is detected, an automated alert will be sent to study staff via email or SMS to prompt immediate intervention. In addition, all participants will receive treatment as usual.

DETAILED DESCRIPTION:
This study will employ a multi-site, single-arm design. A total of approximately 50-100 participants - patients stable for at least 2 weeks on their current opioid replacement medication - will be recruited for the study. All participants will receive their doctor's treatment-as-usual. Patients not currently prescribed Zubsolv® will be switched to Zubsolv®.

Study visits include a screening visit, one baseline visit (which ideally will occur between 7 and 14 days after the screening visit), and bi-weekly visits for the 12 weeks (six visits) following the baseline visit. During the baseline visit, participants will be trained on how to use the AiCure app. Training consists of a number of interactive training steps to teach the participant how to use the app correctly. Participants will be provided with three placebo tablets for the training.

Study participants will be reimbursed to cover their time and transportation costs in accordance with Institutional Review Board (IRB) guidelines. Participants will receive contingency management (CM) to reinforce regular use of the app. Orexo AB will provide the study drug, Zubsolv®, to all participants throughout the 12-week treatment duration.

For the length of the study, participants will be requested to take each dose of their prescribed Zubsolv® regimen using the AiCure app. Each medication administration event will be saved onto the participant's smartphone and encrypted data (including de-identified video and time and date of administration) will be automatically transmitted to the centralized dashboard. Research staff will have access to the dashboard to view real-time and detailed dosing histories for each participant. Access to the dashboard is roles-based and password-protected. If a participant does not dose using the AiCure app (misses/skips a dose), self-reports on the device or over the phone, or is tagged for suspicious behavior, the participant will receive a combination of automated SMS text messages and tailored SMS text messages / phone calls from research staff based on the pre-defined escalation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female at least 18 years of age.
* Has been on a stable dose of buprenorphine/naloxone for at least 2 weeks.
* Is willing to sign a consent form to allow research staff to receive information from their healthcare provider that will verify above inclusion criteria (length of time on stable dose), to administer blood draws, and to perform diagnostic assessments as described in this protocol.
* Is willing to sign an agreement to return the AiCure provisioned device if not able to download AiCure app onto personal smartphone.
* Is willing to use the AiCure app properly each time they ingest their daily dose of buprenorphine/naloxone.
* Is willing to allow research staff (and good clinical practice-trained AiCure personnel) to contact them via the app or other specified means regarding issues related to medication non-adherence.
* Speaks and understands English well enough to participate in the informed consent process and the study assessments and procedures.
* Agrees to come for a research visit monthly for 12 weeks (three visits) after being accepted into the study and two times during screening/baseline.

Exclusion Criteria:

* Is unlikely to remain under the care of their healthcare provider for the duration of the study.
* Appears to be incapable of learning the AiCure system.
* In the opinion of the investigator, is someone who should not be part of the study due to behavioral, mental, physical, or other issues.
* Is under court mandate to obtain treatment.
* Has a known allergy to any of the substances comprising the study medication.
* Is planning to be detoxified from Zubzolv during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and acceptability to participants and study staff in using AiCure to monitor medication adherence. | 12 weeks
  Participants and study staff using AiCure to monitor medication adherence will show high rates of physician satisfaction and user acceptance, based on a pre-post design using surveys and observations.

SECONDARY OUTCOMES:
To evaluate the acceptability of using AiCure to optimize care pathways. | 12 weeks
  Optimization of care pathways will be measured by assessing the sustainability of AiCure use over 12 weeks (retention rates) and measuring the fraction of bi-weekly urines positive for illicit opioids (urine drug screens) compared to historical data.
To measure the reliability and validity of AiCure in detecting interruptions in treatment. | 12 weeks
  Comparing the sensitivity of AiCure adherence data and pharmacokinetic data in detecting interruptions in treatment.
The degree of participant maximum craving (during the 24 hour period prior to the study visit) for opioids as measured by the Brief Substance Craving Scale (BSCS). | 12 weeks
The change in participant's psychosocial well being over time as measured by the seven subscales of the Addiction Severity Index (ASI). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alain Litwin, MD, Principal Investigator — Montefiore Medical Center; Adam Hanina, MBA, MPhil, Study Director — AiCure
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No